CLINICAL TRIAL: NCT03591588
Title: Effects of Diet Interventions on Monocyte Phenotypes in Individuals With Metabolic Syndrome
Brief Title: Effects of Diet Interventions on Monocytes in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Huaizhu Wu, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H21418
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Metabolic Syndrome; Hypertriglyceridemia
MeSH Terms: conditions — Metabolic Syndrome; Hypertriglyceridemia | interventions — Diet

STUDY DESIGN:
Intervention Model Description: The study includes 2 types of diets, i.e., high-saturated fat diet and low-fat high-protein diet, in the same individuals with randomized crossover design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-saturated fat diet (Active Comparator): Diet high in saturated fat (~50% calorie from fat, ~25% from saturated fat)
  Interventions: Other: diet
- low-fat diet (Active Comparator): Diet with low fat (~25% calorie from fat)
  Interventions: Other: diet

INTERVENTIONS:
Other: diet — The study includes 2 types of diets, i.e., high-saturated fat diet and low-fat high-protein diet, which are provided to each participant in a randomized crossover design.

SUMMARY:
Subjects with hypertriglyceridemia and metabolic syndrome are being recruited and receive diet interventions with either a high-saturated fat diet or a low-fat high protein diet for 4 days (days 1-4) and a breakfast on day 5. Blood samples are collected on day 1 and day 5 to examine lipid levels and circulating monocyte phenotypes.

DETAILED DESCRIPTION:
Subjects with hypertriglyceridemia and metabolic syndrome are being recruited and receive diet interventions with either a high-saturated fat diet or a low-fat high protein diet for 4 days (days 1-4) and a breakfast on day 5. Blood samples are collected on day 1 at fasting state and on day 5 at fasting state and 4 and 6 hours after the breakfast to examine lipid levels and circulating monocyte phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Obese women and men with metabolic syndrome (MS)
* Fasting triglyceride (TG) equal to or greater than 150 mg/dl

Exclusion Criteria:

* <21 years of age
* Perimenopausal, pregnant or breastfeeding women
* Current smokers
* Obvious inflammation or other acute illnesses
* Obesity due to endocrinologic disorders including polycystic ovary syndrome
* Partial lipodystrophy
* Diabetes requiring insulin or >1 oral medication
* Fasting TG ≥650 mg/dl
* A history of pancreatitis
* Myocardial infarction within the past 3 years
* Any hospitalization within the past 2 months
* Takes steroids.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Effects of diet interventions on monocyte phenotypes | 2016 to 2020
  Monocyte phenotypes

CONTACTS AND LOCATIONS:
Overall Officials: HUAIZHU WU, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Center for Prevention of cardiometabolic disease, Houston, Texas, United States

REFERENCES:
- [Derived] Lian Z, Perrard XD, Antony AK, Peng X, Xu L, Ni J, Zhang B, O'Brien V, Saeed A, Jia X, Hussain A, Yu B, Simon SI, Sacks FM, Hoogeveen RC, Ballantyne CM, Wu H. Dietary Effects on Monocyte Phenotypes in Subjects With Hypertriglyceridemia and Metabolic Syndrome. JACC Basic Transl Sci. 2023 Apr 26;8(5):460-475. doi: 10.1016/j.jacbts.2023.02.011. eCollection 2023 May. PMID 37325398